CLINICAL TRIAL: NCT00584922
Title: Early Detection and Treatment of Esophageal Injury After Catheter Ablation for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 13165
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation
Keywords: Esophageal injury; Catheter Ablation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AF ablation group: Patients undergoing catheter ablation of atrial fibrillation or left atrial macroreentrant tachycardia.
  Interventions: Procedure: Endoscopy in group I (all patients)

INTERVENTIONS:
Procedure: Endoscopy in group I (all patients) — Post procedure endoscopy, omeprazole 40 mg BID, sucralfate 1 gm BID for 2-4 weeks.

SUMMARY:
The purpose of this study is to prospectively follow the next 200 patients who undergo catheter ablation of atrial fibrillation for symptoms and signs of esophageal injury.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively follow the next 200 patients who undergo catheter ablation of atrial fibrillation and endoscopy. If any signs of esophageal injury are seen on endoscopy the patients will be treated with omeprazole and sucralfate and they will have repeat endoscopy in two weeks. Patients who do not have any esophageal injury will be contacted by telephone in two weeks to be assessed for GI symptoms.

Specific Aims: The specific aims of the study are to:

1. Assess the incidence of visible transmural esophageal injury following extensive ablation in the posterior left atrium as measured by endoscopy1
2. Assess whether early detection of esophageal injury by endoscopy and treatment will prevent development of more serious injury such as left atrial-esophageal fistula
3. Identify predictors of esophageal injury. In particular, to assess if esophageal temperature rises during ablation correlate with development of esophageal injury and if the absence of esophageal temperature rise during ablation correlate with the absence of esophageal injury.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Scheduled to have catheter ablation of atrial fibrillation or left atrial macroreentrant tachycardia.

Exclusion Criteria:

* Contraindication to endoscopy
* Pregnancy
* Prisoners
* Inability or unwillingness to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-80 scheduled to undergo catheter ablation of atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2006-12-05 (Actual); Primary Completion 2011-03-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Beckman, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AF Ablation Group
Started | 175
Completed | 175
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AF Ablation Group
Number analyzed (Participants) | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 131
  >=65 years | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 140
Region of Enrollment [Number; unit: participants]
  United States | 175

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Esophageal Injury as Assessed by Endoscopy
Description: Endoscopy results and clinical status at one month after endoscopy procedure.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | AF Ablation Group
Number analyzed (Participants) | 175
participants
  Erythema | 1
  Erosion | 12
  Ulcer | 4
  Fistula | 0
  None | 158

ADVERSE EVENTS:
Time Frame: Endoscopy one day after ablation Clinical evaluation 1 month after ablation
Description: Adverse events were collected by:
  1. endoscopy results
  2. Telephone survey at one month
Arm/Group | AF Ablation Group
All-Cause Mortality (participants affected / at risk) | 0/171
Serious Adverse Events (participants affected / at risk) | 17/171
Other Adverse Events (participants affected / at risk) | 0/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AF Ablation Group (N=171)
Esophageal erythema (Gastrointestinal disorders) | 1 (1) — by endoscopy
Esophageal erosion (Gastrointestinal disorders) | 12 (12) — by endoscopy
Esophageal Ulcer (Gastrointestinal disorders) | 4 (4) — By endoscopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes